CLINICAL TRIAL: NCT01632969
Title: Improving End of Life Care in Head and Neck Cancer
Status: Terminated | Type: Observational
Why Stopped: Lack of accrual
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 12-136
Record Dates: First submitted 2012-06-29; First posted 2012-07-04 (Estimated); Last update posted 2015-03-06 (Estimated); Status verified 2015-03

CONDITIONS: The Families or Next of Kin of Patients Treated at MSKCC for Non-cutaneous Squamous Cell Carcinomas of the; Upper Aerodigestive Tract
Keywords: 12-136
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- families or next-of-kin of deceased patients: The families of deceased patients treated at MSKCC for non-cutaneous squamous cell carcinomas of the upper aerodigestive tract for whom contact information is available will be recruited by mail and by phone.
  Interventions: Behavioral: The The Family Assessment of Treatment at the End of life (FATE ) survey

INTERVENTIONS:
Behavioral: The The Family Assessment of Treatment at the End of life (FATE ) survey — Study candidates will be contacted by mail with an initial contact letter with information explaining the study, and then will receive a follow-up phone call to discuss their participation in the study no later than 1 month following the posting of the initial contact letter. If a family member or next-of-kin chooses to participate, verbal informed consent will be obtained over the phone and a one-time telephone interview will be conducted.

SUMMARY:
The purpose of this study is to improve the quality of care provided for head and neck cancer patients. By better understanding the end of life experiences of dying patients and their families, the investigators hope to better anticipate and improve upon the experiences of future patients and their families.

ELIGIBILITY:
Inclusion Criteria:

* Head and neck cancer patients who received their treatment at MSKCC who have died of noncutaneous squamous cell carcinomas of the upper aerodigestive tract and for whom family / next of kin contact information is available.
* Time of patient death must have been at least 6 months ago and no more than 4 years ago
* Patient age at time of death must be over 21 years of age.
* Those interviewed must be English-fluent.

Exclusion Criteria:

* Non-English speaking interviewees
* Next-of-kin who reported being unfamiliar with care received during the last month of life
* Next-of-kin who did not identify themselves as one of the patient's primary social supports during the last month of life
* Next-of-kin who were not physically present with the deceased at least once during the last week of his/her life
* Next-of-kin under age 21

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Deceased Head and Neck Surgery patients will be queried from Dataline and screened for eligibility. Interviews with family members and next of kin of deceased patients treated at MSKCC for noncutaneous squamous cell carcinomas of the upper aerodigestive tract will be conducted via telephone, employing the survey instruments.
Sampling Method: Non-Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2012-06; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
quality of care received by patients | 1 year
  To determine the perception of the family members of the quality of care received by patients with aerodigestive mucosal squamous cell carcinoma of the head and neck at the end of their lives. A survey will be administered to the families and next-of-kin of deceased patients. A recently validated survey instrument, the Family Assessment of Treatment at the End of life (FATE), is designed to assess treatment at the end of life based upon the responses of family members of the deceased (Finlay, Shreve et al. 2008).

SECONDARY OUTCOMES:
quality of death outcomes | 1 year
  To identify specific risk factors or interventions that might predict certain quality of death outcomes. A survey will be administered to the families and next-of-kin of deceased patients.A recently validated survey instrument, the Family Assessment of Treatment at the End of life (FATE), is designed to assess treatment at the end of life based upon the responses of family members of the deceased (Finlay, Shreve et al. 2008).
awareness among caregivers | 1 year
  To raise awareness among caregivers of the perspectives of family members of deceased patients, and of risk factors that might predict patient quality of death. This survey will be administered to the families and next-of-kin of deceased patients. A recently validated survey instrument, the Family Assessment of Treatment at the End of life (FATE), is designed to assess treatment at the end of life based upon the responses of family members of the deceased (Finlay, Shreve et al. 2008).

CONTACTS AND LOCATIONS:
Overall Officials: Snehal Patel, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/